CLINICAL TRIAL: NCT04422925
Title: In Living Donor Hepatectomy Cases, the Preoperative and Postoperative Relationship Between s100β, NSE and GFAP Levels and Postoperative Delirium
Brief Title: s100β, NSE n GFAP in Living Donor Hepatectomy and Delirium
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Bora Dinc, MD. Assist. Prof., Akdeniz University
Other Study IDs: s100β, NSE n GFAP in LDH
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Donor Site Complication; Delirium; Uremic Encephalopathy; Neurologic Manifestations
Keywords: donor living hepatectomy; s100β; neuron specific enolase; glial fibrillary acidic protein; delirium
MeSH Terms: conditions — Delirium; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — s100β, neuron specific enolase and glial fibrillary acidic
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Living Donor Hepatectomy — On living donor hepatectomy (preoperative), the first following day of surgery, 3rd day, and 7th day, blood will be taken for the measurement of S100β, NSE, and GFAP levels in the postoperative period. The plasma of the blood taken will be separated and stored at -800C. Values will be measured by the ELISA method. During the hospitalization, the delirium status of the patients will be evaluated with the delirium evaluation scale (Delirium Rating Scale-Revised - 98 Turkish version). Functional and cognitive information and other results will be collected at each follow-up point.

SUMMARY:
The post-operative delirium picture is a serious and common complication seen after any major surgery, including hepatic resection. Patients who will be planned to undergo donor hepatectomy for liver transplantation will be included in the study. Basic clinical and demographic information of patients undergoes donor hepatectomy will be recorded before surgery. The anatomical parameters such as liver volume, medications performed during the surgery, complications, bleeding amounts, fluids given, blood and blood products, vital signs during surgery, fluid balance, duration of surgery, recovery length at post-operative period, complications after surgery, approaches to complications, analgesics and other medications used, hemogram and other biochemical parameters (electrolytes, albumin, liver frontier tests, etc.), weight status, vital signs, duration of intensive care, post-operative VAS scores, drainage and information such as length of stay, length of hospital stay, the healing time of the wound will also be recorded.

During the hospitalization, the delirium status of the patients will be evaluated with a delirium evaluation scale by consultant doctor. Blood will be taken for the measurement of S100β, NSE, and GFAP levels one day before donor hepatectomy and following day of hepatectomy, 3rd day, and 7th day in the post-operative period. The plasma of the blood taken will be separated and stored at -80 0C until working. Laboratory values are taken from the patients before the operation will be recorded over the system. The relationship between the results obtained and the delirium evaluation scores performed on the days followed will be evaluated.

This study aims to analyze the delirium incidence and post-operative early S100β, NSE, and GFAP levels within the first week following the hepatectomy performed in live donors for liver transplantation.

DETAILED DESCRIPTION:
The postoperative delirium picture is a serious and common complication seen after any major surgery, including hepatic resection. Delirium is an acute state of confusion characterized by impaired consciousness, reduced ability to focus on attention, changes in cognitive functions, a perceptual disturbance development, and an uncomfortable sleep-wake cycle. Postoperative delirium has an acute onset and has a fluctuating course. This complication results in a long recovery period, a longer stay in the intensive care unit, higher complication rates, extra nursing care, and higher costs. Therefore, appropriate methods are needed to prevent and treat postoperative delirium.

The pathophysiology of delirium is thought to be due to many reasons. Examined in titles: Changes in the electrolyte and fluid balance, nutritional imbalance (low serum protein/albumin level, hypovitaminosis, especially cobalamin deficiencies (B12), folate (B9), niacin (B3, pellagra), thiamine, age (> 65) and gender (m> f), hyperthermia and hypothermia, major surgical procedures, endocrine disorders, drug use, anemia, anoxia, hypoxia and low perfusion/oxygenation states, postoperative pain and painkiller medication, end-organ failure, social isolation, decreased intellectual stimulation (long-term intensive care therapy), sleep disorders and changes in the circadian rhythm, metabolic disorders (acidosis, alkalosis, hyperammonemia, hypersensitivity reactions, glucose, and acid-base disorders, limitations, and inactivity. Cases are exposed to these predisposing causes.

Postoperative delirium is a type of delirium that is exposed to surgical procedure and anesthesia, usually seen between the 1st and 3rd days after surgery. Postoperative delirium can be seen at rates ranging from 9 to 87% depending on the age of the patient and the type of surgery. Although its etiology is not yet understood, it is probably thought to be multifactorial.

S100β is secreted by astrocytes in brain damage. S100β rises while brain damage starts, so it can be used in the diagnosis of early brain damage. Neuron-specific enolase (NSE) acts as an intracytoplasmic enzyme, and serum levels are increased in neuron damage. The glial fibrillar acidic protein (GFAP) is the intermediate filament cytoskeleton protein in astrocytes. It originates from the same root structure as S100β. After hepatectomy, the donor candidates are exposed to physiological changes that include the central nervous system due to surgical stress as well as the functional change of the remaining liver tissue. Determining the increase in serum level of biomarkers specific to the central nervous system mentioned before the development of cognitive disorders such as delirium may prevent the complications that may arise during the postoperative period. It also helps to provide treatment in the postoperative period as well as evaluation.

The aim of this study is to analyze the delirium incidence and postoperative early S100β, NSE, and GFAP levels within the first week following the hepatectomy performed in living donors for liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are admitted as a donor who will undergo living donor hepatectomy operation by Akdeniz University Faculty of Medicine Organ Transplant Center and planned to have a donor right hepatectomy operation
* Patients who have read and accepted the detailed informed consent form

Exclusion Criteria:

* Failure to supply routine blood sampling during follow-up
* Having major complications after surgery (pulmonary embolization, sepsis, etc.)
* Individuals with mental health disorders detected by the organ transplantation committee in the preoperative period.

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients' demographic data (age, gender, weight, height), accompanying diseases, ASA classification, main etiology, preoperative serums taken in the preoperative period; serum sodium, potassium, ammonium, total bilirubin, ALT, AST, albumin, alkaline phosphatase, INR, creatinine, and BUN shall be recorded accordingly. In addition, routinely taken anesthetics, duration of the operation, duration of anesthesia, duration before the reperfusion, duration of postperfusion, first measured central venous pressure, volume replacement therapy, blood component transfusion, the total fluid amount given during the operation, corticosteroids and immunosuppressive drugs given during the operation shall be recorded. Besides, the cognitive functions of the patients and blood samples for mentioned values will be evaluated in the preoperative and postoperative periods.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Assessment of serum s100β | 2 years
  Approximately 25 patients planned to have living donor hepatectomy will be included in the study. The blood samples are taken in the preoperative period before the induction of anesthesia in the operating room and postoperative (the first day, the third day and the seventh day) period to analyze S100β serum concentrations and neurologic damage of living donor hepatectomy patients besides evaluating its effect on prognosis. These samples shall be kept at -80 0C until the plasma separation process.
Assessment of serum NSE | 2 years
  Approximately 25 patients planned to have living donor hepatectomy will be included in the study. The blood samples are taken in the preoperative period before the induction of anesthesia in the operating room and postoperative (the first day, the third day and the seventh day) period to analyze NSE serum concentrations and neurologic damage of living donor hepatectomy patients besides evaluating its effect on prognosis. These samples shall be kept at -80 0C until the plasma separation process.
Assessment of serum GFAP | 2 years
  Approximately 25 patients planned to have living donor hepatectomy will be included in the study. The blood samples are taken in the preoperative period before the induction of anesthesia in the operating room and postoperative (the first day, the third day and the seventh day) period to analyze GFAP serum concentrations and neurologic damage of living donor hepatectomy patients besides evaluating its effect on prognosis. These samples shall be kept at -80 0C until the plasma separation process.
Assessment of serum cognitive functions and delirium status | 2 years
  During the hospitalization, the delirium status of the patients will be evaluated with the delirium evaluation scale (Delirium Rating Scale-Revised - 98 Turkish version). Functional and cognitive information and other results will be collected at each follow-up point.

CONTACTS AND LOCATIONS:
Overall Officials: Bora Di̇nc, MD, Assist. Prof., Study Director — Akdeniz University Medical Faculty
Locations (1):
- Akdeniz University Medical Faculty Department of Anesthesiology and Reanimation, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided